CLINICAL TRIAL: NCT04898140
Title: The Evaluation of the Intensity of Cellular and Humoral Immunity to COVID-19 Causative Agent in Moscow Residents
Brief Title: The Evaluation of Cellular and Humoral Immunity to COVID-19 in Moscow Residents
Status: Completed | Type: Observational
Sponsor: Moscow Department of Health (Other Government)
Collaborators: Clinical City Hospital named after I.V. Davydovsky of Moscow Department of Healthcare (Network); Moscow State University of Medicine and Dentistry (Other); Moscow Institute of Physics and Technology (Unknown); National Research Center for Hematology, Russia (Network); State Research Center Institute of Immunology, Russia (Unknown); Shemyakin-Ovchinnikov Institute of bioorganic chemistry RAS (Unknown); National Medical Research Center of Phthisiopulmonology and Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1027739482649/0908/4_9
Record Dates: First submitted 2021-05-21; First posted 2021-05-24 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Covid19; Respiratory Viral Infection
Keywords: Covid19; T cell immunity; virus-specific antibodies; protective immunity; flow cytometry; ELISpot
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood plasma and serum. Peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy volunteers: Individuals who were not infected and not having been demonstrated COVID-19 symptoms since December 2019.
  Interventions: Diagnostic Test: SARS-CoV-2 specific IgM and IgG detection; Diagnostic Test: ELISpot: detection of the T cells specific to different SARS-CoV-2 proteins; Diagnostic Test: Flow cytometry: detection of the SARS-CoV-2 specific T-helpers and cytotoxic T lymphocytes
- Recovered: Individuals who were recovered from COVID-19 with different severity.
  Interventions: Diagnostic Test: SARS-CoV-2 specific IgM and IgG detection; Diagnostic Test: ELISpot: detection of the T cells specific to different SARS-CoV-2 proteins; Diagnostic Test: Flow cytometry: detection of the SARS-CoV-2 specific T-helpers and cytotoxic T lymphocytes
- Vaccinated: Individuals who were vaccinated against SARS-CoV-2 with "Sputnik V" vaccine.
  Interventions: Diagnostic Test: SARS-CoV-2 specific IgM and IgG detection; Diagnostic Test: ELISpot: detection of the T cells specific to different SARS-CoV-2 proteins; Diagnostic Test: Flow cytometry: detection of the SARS-CoV-2 specific T-helpers and cytotoxic T lymphocytes
- Special group: Individuals who recovered from COVID-19 concomitant with other immune-related comorbidities (tuberculosis, chronic obstructive pulmonary disease, HIV infection, hematological neoplasia).
  Interventions: Diagnostic Test: SARS-CoV-2 specific IgM and IgG detection; Diagnostic Test: ELISpot: detection of the T cells specific to different SARS-CoV-2 proteins; Diagnostic Test: Flow cytometry: detection of the SARS-CoV-2 specific T-helpers and cytotoxic T lymphocytes

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 specific IgM and IgG detection — Detection of IgM and IgG antibodies specific to the SARS-CoV-2 antigens in the blood serum using enzyme-linked immunosorbent assay (ELISA).
Diagnostic Test: ELISpot: detection of the T cells specific to different SARS-CoV-2 proteins — Detection of peripheral blood T lymphocytes which are activated and secrete interferon gamma (IFNgamma) upon stimulation with peptides, covering the immunodominant sequence domains of the nucleocapsid N, membrane M, or spike glycoprotein S proteins of SARS-CoV-2 coronavirus.
Diagnostic Test: Flow cytometry: detection of the SARS-CoV-2 specific T-helpers and cytotoxic T lymphocytes — Detection of peripheral blood T-helpers (CD45+CD3+CD4+)* and cytotoxic T cells (CD45+CD3+CD8+)* which are activated and secrete IFNgamma and/or interleukin-2 (IL2) upon stimulation with mixture of peptides, covering the immunodominant sequence domains of the nucleocapsid N, membrane M, and spike glycoprotein S proteins of SARS-CoV-2 coronavirus. * CD, cluster of differentiation

SUMMARY:
The aim of the research is to estimate the levels of cellular and humoral immunity to the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) among Moscow residents over 18 years old. During the study, participants will be divided into four groups: healthy volunteers; individuals recovered from coronavirus disease 2019 (COVID-19) with different severity; individuals vaccinated against SARS-CoV-2; individuals who have had COVID-19 concomitantly with comorbidities that characterized by the impact on the immune system (tuberculosis, chronic obstructive pulmonary disease, HIV infection, hematological neoplasia). For all participants included into the study peripheral blood will be collected and the titers of SARS-CoV-2 specific immunoglobulins M (IgM) and immunoglobulins G (IgG), frequencies of the T cells specific to nucleocapsid (N), membrane (M), and spike (S) proteins of SARS-CoV-2 in peripheral blood, as well as the fractions of virus specific T helpers and cytotoxic T cells will be estimated. For smaller cohorts of the participants in all groups the antibody titers and T cell response levels will be examined in dynamics. All participants will be monitored for the incidence of primary or repeated COVID-19 for 1-2 years after inclusion in the study.

Based on the results of the study, the relationship between the formation of humoral and cellular immunity against COVID-19, the duration of these types of immunity, as well as their individual contribution to protection against primary or secondary SARS-CoV-2 infection will be analyzed. Additionally, data concerning patients recovered from COVID-19 and having concomitant diseases will provide a valuable information that may help to understand in more details the mechanisms of the development of the SARS-CoV-2 specific immune response.

ELIGIBILITY:
Inclusion Criteria:

* residents of the Moscow city (registered in Moscow);
* 18 years old or above;
* signed informed consent.

Exclusion Criteria:

* citizenship of a foreign state;
* refusal to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Moscow city over 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 5340 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
IgM/IgG titer | At the moment of inclusion and for 1-2 years after inclusion in the study.
  The level of SARS-CoV-2 specific IgM/IgG antibodies in blood serum.
Peripheral blood T cells specific to different SARS-CoV-2 proteins | At the moment of inclusion and for 1-2 years after inclusion in the study.
  The number of peripheral blood T cells specific to N, M or S protein of SARS-CoV-2.
Subpopulations of SARS-CoV-2 specific peripheral blood T lymphocytes | At the moment of inclusion and for 1-2 years after inclusion in the study.
  The number of peripheral blood T-helpers and cytotoxic T cells specific to SARS-CoV-2 coronavirus antigens.
Primary or repeated COVID-19 cases | 1-2 years after inclusion in the study.
  Monitoring of the SARS-CoV-2 infection cases, severity of symptoms, outcomes and recovery period among participants included into the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical City Hospital named after I.V. Davydovsky of Moscow Department of Healthcare, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Molodtsov IA, Kegeles E, Mitin AN, Mityaeva O, Musatova OE, Panova AE, Pashenkov MV, Peshkova IO, Alsalloum A, Asaad W, Budikhina AS, Deryabin AS, Dolzhikova IV, Filimonova IN, Gracheva AN, Ivanova OI, Kizilova A, Komogorova VV, Komova A, Kompantseva NI, Kucheryavykh E, Lagutkin Dcapital A, Cyrillic, Lomakin YA, Maleeva AV, Maryukhnich EV, Mohammad A, Murugin VV, Murugina NE, Navoikova A, Nikonova MF, Ovchinnikova LA, Panarina Y, Pinegina NV, Potashnikova DM, Romanova EV, Saidova AA, Sakr N, Samoilova AG, Serdyuk Y, Shakirova NT, Sharova NI, Sheetikov SA, Shemetova AF, Shevkova LV, Shpektor AV, Trufanova A, Tvorogova AV, Ukrainskaya VM, Vinokurov AS, Vorobyeva DA, Zornikova KV, Efimov GA, Khaitov MR, Kofiadi IA, Komissarov AA, Logunov DY, Naigovzina NB, Rubtsov YP, Vasilyeva IA, Volchkov P, Vasilieva E. Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)-Specific T Cells and Antibodies in Coronavirus Disease 2019 (COVID-19) Protection: A Prospective Study. Clin Infect Dis. 2022 Aug 24;75(1):e1-e9. doi: 10.1093/cid/ciac278. PMID 35435222
- [Result] Komissarov AA, Dolzhikova IV, Efimov GA, Logunov DY, Mityaeva O, Molodtsov IA, Naigovzina NB, Peshkova IO, Shcheblyakov DV, Volchkov P, Gintsburg AL, Vasilieva E. Boosting of the SARS-CoV-2-Specific Immune Response after Vaccination with Single-Dose Sputnik Light Vaccine. J Immunol. 2022 Mar 1;208(5):1139-1145. doi: 10.4049/jimmunol.2101052. Epub 2022 Jan 31. PMID 35101893
- See also: Official website of Clinical City Hospital named after I.V. Davydovsky of Moscow Department of Healthcare — http://gkb-23.ru